CLINICAL TRIAL: NCT03867500
Title: Effects of Niacin on Intramyocellular Fatty Acid Trafficking in Upper Body Obesity and Type 2 Diabetes Mellitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principle Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17-009977; 5R01DK045343 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-03-08 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Niacin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niacin then saline (Experimental): All participants will receive intravenous Niacin overnight on day one and then intravenous saline overnight on the second study day
  Interventions: Drug: Niacin; Drug: Saline

INTERVENTIONS:
Drug: Niacin — Intravenous infusion, a titrated dose starting from 0.6 mg/min to a maximum of 2.8 mg/min (likely needed dose = 1.4 mg/min)
Drug: Saline — Intravenous infusion of 0.9% Sodium chloride (NaCl)

SUMMARY:
Muscle insulin resistance is a hallmark of upper body obesity (UBO) and Type 2 diabetes (T2DM). It is unknown whether muscle free fatty acid (FFA) availability or intramyocellular fatty acid trafficking is responsible for the abnormal response to insulin. Likewise, the investigators do not understand to what extent the incorporation of FFA into ceramides or diacylglycerols (DG) affect insulin signaling and muscle glucose uptake. The investigators will measure muscle FFA storage into intramyocellular triglyceride, intramyocellular fatty acid trafficking, activation of the insulin signaling pathway and glucose disposal rates under both saline control (high overnight FFA) and after an overnight infusion of intravenous niacin (lower/normal FFA) to provide the first integrated examination of the interaction between FFA and muscle insulin action from the whole body to the cellular/molecular level. By identifying which steps in the insulin signaling pathway are most affected, the investigators will determine the site-specific effect of ceramides and/or DG on different degrees of insulin resistance.

Hypothesis 1: Greater trafficking of plasma FFA into intramyocellular DG will impair proximal insulin signaling and reduce muscle glucose uptake.

Hypothesis 2: Lowering FFA in UBO and T2DM by using an intravenous infusion of niacin will alter trafficking of plasma FFA into intramyocellular ceramides in a way that will improve insulin signaling and increase muscle glucose uptake.

Hypothesis 3: Lowering FFA in UBO and T2DM by using an intravenous infusion of niacin will alter trafficking of plasma FFA into intramyocellular DG in a way that will improve insulin signaling and increase muscle glucose uptake.

ELIGIBILITY:
Inclusion criteria:

* Women and Men (Women premenopausal)
* BMI 29-37
* Weight stable
* Not pregnant/nursing

Exclusion criteria:

* Ischemic heart disease
* Atherosclerotic valvular disease
* Smokers (>20 cigarettes per week)
* Bilateral oophorectomy
* Concomitant use of medications that can alter serum lipid profile:

  * High dose fish oil (>3g per day),
  * STATINS (if yes hold for 6 weeks and receive PCP's approval),
  * Niacin
  * Fibrates
  * thiazolidinediones
  * Beta-blockers
  * Atypical antipsychotics
* Lidocaine or Niacin/Niaspan allergy
* Subjects with 1.5 times upper limit of normal of serum creatinine, Alkaline phosphatase, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) unless participant has fatty liver disease, Total bilirubin (unless the patient has documented Gilbert's syndrome)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Niacin Then Saline: Participants received intravenous Niacin overnight on day one and then intravenous saline overnight on the second study day
  Niacin: Intravenous infusion, a titrated dose starting from 0.6 mg/min to a maximum of 2.8 mg/min (likely needed dose = 1.4 mg/min)
  Saline: Intravenous infusion of 0.9% Sodium chloride (NaCl)
Period: Niacin Infusion Intervention
Arm/Group | Niacin Then Saline
Started | 12
Completed | 12
Not Completed | 0
Period: Saline Infustion Intervention
Arm/Group | Niacin Then Saline
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Niacin Then Saline
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Glucose Infusion Rate
Description: Glucose infusion rates will be measured in upper body obese and type 2 diabetic volunteers using hyperinsulinemic, euglycemic clamp under saline control conditions and during an intravenous infusion of niacin. The hyperinsulinemic-euglycemic clamp is a method used to measure insulin sensitivity. Plasma insulin concentration is acutely raised and maintained at ~40-80 μU/ml (microunits per milliliter) by continuous insulin infusion. During the clamp, the plasma glucose concentration was held constant at normal blood sugar level. The glucose infusion rate over the last hour of the insulin infusion is the net effect of insulin on whole-body glucose metabolism. This rate serves as a measure of tissue insulin sensitivity. The hyperinsulinemic-euglycemic clamp assesses how sensitive your tissues are to insulin.
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: microunits per milliliter
Groups:
- Niacin: Participants who received intravenous Niacin overnight on day one
  Niacin: Intravenous infusion, a titrated dose starting from 0.6 mg/min to a maximum of 2.8 mg/min (likely needed dose = 1.4 mg/min)
- Saline: Participants who received intravenous saline overnight on the second study day
  Saline: Intravenous infusion of 0.9% Sodium chloride (NaCl)
Arm/Group | Niacin | Saline
Number analyzed (Participants) | 11 | 11
microunits per milliliter | 532 (214) | 557 (256)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline, first intervention of Niacin, second intervention of Saline to end of study, approximately eight weeks
Arm/Group | Niacin | Saline
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin (N=12) | Saline (N=11)
muscle biopsy discomfort or drainage (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Bloody or non-bloody drainage at the site of muscle biopsy or discomfort that involved physician assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03867500/Prot_SAP_000.pdf